CLINICAL TRIAL: NCT06466083
Title: Correlation Analysis of Postoperative Delirium and Postoperative Neurocognitive Disorder in Elderly Spinal Surgery Patients
Brief Title: Correlation Analysis of POD and pNCD in Elderly Spinal Surgery Patients
Status: Recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: 19880416
Record Dates: First submitted 2024-05-29; First posted 2024-06-20 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Delirium; Postoperative Neurocognitive Disorder; Spinal Surgery
Keywords: postoperative delirium; postoperative neurocognitive disorder; serum indexes; spinal surgery
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- postoperative delirium(POD) and postoperative neurocognitive disorder(pNCD): Delirium (CAM scale ) was assessed 7 days after surgery and divided into POD and non-POD groups; one of the above scenarios indicated postoperative delirium;The patients in the POD group were evaluated for cognitive function at 1 month and 12 months after surgery to determine whether pNCD occurred. The patients in the POD group were further divided into pNCD subgroup and non-PNCD subgroup, and serum indexes were compared
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — this is an observation study,no intervention

SUMMARY:
This study is a prospective cohort study to investigate the differences in serum indexes between elderly spinal surgery patients with postoperative delirium (POD) who either develop or do not develop long-term postoperative neurocognitive disorders (pNCD).

DETAILED DESCRIPTION:
To investigate the differences in serum indexes between elderly spinal surgery patients with postoperative delirium (POD) who either develop or do not develop long-term postoperative neurocognitive disorders (pNCD).

Neurocognitive function of the study participants was assessed within one week before surgery using the Montreal Cognitive Assessment (MoCA). Compare changes in serum indexes level before and after surgery. Under routine anesthetic management of the Department of Anesthesiology and Surgical Operations at Xuanwu Hospital, endotracheal intubation general anesthesia was performed. Within 7 days post-surgery, delirium assessment was conducted using the Confusion Assessment Method (CAM), classifying patients into POD and non-POD groups. Neurocognitive function assessments were conducted long-term after surgery for the POD group to determine the presence of pNCD, further dividing the POD group into pNCD and non-pNCD subgroups, followed by serum indexes.By comparing the changes of serum indexes before and after surgery between the pNCD and non-pNCD subgroups, exploring the correlation of POD and pNCD.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥65 years of age who have undergone spinal surgery anesthesia; Sign informed consent

Exclusion Criteria:

* Inability to complete cognitive function assessment; Illiteracy, hearing impairment or visual impairment; He has a history of epilepsy, depression, schizophrenia, Alzheimer's disease and other psychiatric and neurological diseases

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients 65~100 years of age who have undergone spinal surgical anesthesia
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2025-01-14 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
change in serum indexes between elderly spinal patients with postoperative delirium(POD) who either develop or do not develop postoperative neurocognitive disorders (pNCD) one month after surgery | 2024.5.9-2026.5.1
  Perioperative neurocognitive disorders (PND) represent one of the common complications of general anesthesia, posing serious hazards and currently being a hot topic and a challenging problem in international research. Recently, general anesthesia has led to a new breakthrough in the study of PND serum-related markers, such as brain-derived nutritional factors(BDNF)、C-reactive protein(CRP)、homocysteine(Hcy). This provides new perspectives for PND prevention, evaluation and furnishes theoretical grounds for enhancing the safety of clinical anesthesia and the quality of life for patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, 100053, Beijing, China

IPD SHARING:
Plan to Share IPD: No